CLINICAL TRIAL: NCT01932034
Title: Prospective Study to Optimize Vancomycin Dosing in Children and Adults Using Multiple-Model Bayesian Adaptive Control
Brief Title: Prospective Study to Optimize Vancomycin Dosing in Children and Adults Using Computer Software
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Michael Neely, Michael Neely, MD, MSc, FCP, Children's Hospital Los Angeles
Other Study IDs: LACUSC-Van-01; R01GM068968 (NIH)
Record Dates: First submitted 2013-08-06; First posted 2013-08-30 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Bacterial Infections
Keywords: Vancomycin; Pharmacokinetics; Pharmacodynamics; Decision support
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Standard dosing: Vancomycin dosed and monitored according to standard practice
- BestDose Computer Software: Vancomycin dosed using BestDose computer software, targeting AUC rather than trough concentrations
  Interventions: Device: BestDose Computer Software
- BestDose Computer Software 2: Vancomycin dosed using BestDose computer software, targeting AUC rather than trough concentrations and with computer-generated suggested optimal blood sampling times
  Interventions: Device: BestDose Computer Software

INTERVENTIONS:
Device: BestDose Computer Software — BestDose is made by the USC Laboratory of Applied Pharmacokinetics. It uses a multiple-model, Bayesian adaptive control algorithm to find the maximally precise dose that will achieve a user-specified target concentration or concentrations.
  Groups: BestDose Computer Software; BestDose Computer Software 2

SUMMARY:
We will compare the percentage of patients having therapeutic vancomycin serum concentrations after current standard dosing, after dosing with our software. We will also include therapeutic outcomes and costs in the analysis.

DETAILED DESCRIPTION:
Recent guidelines to use the antibiotic vancomycin for serious, resistant gram-positive bacterial infections advocate higher plasma concentrations than are routinely achieved with conventional dosing. Moreover, there is wide interpatient variability in vancomycin plasma concentrations, even with standardized dosing. The hypothesis for this study is that dosing vancomycin assisted by computer software and Bayesian algorithms will lead to more rapid and accurate attainment of therapeutic blood vancomycin concentrations in children and adults. This study will enroll 90 patients per year for three years, totaling 270 patients. Eligible patients will be of any age and who are to be prescribed vancomycin by their clinicians for medical indications. Patients with vancomycin-resistant organisms, severe vancomycin allergies or who need dialysis will not be eligible. Participants in the first group of 90 will be treated according to standard care. The second and third groups of patients will be dosed with vancomycin according to the recommendations made by the study team using the BestDose software developed by the USC Laboratory of Applied Pharmacokinetics. The second group will be dosed with the software in its current form, and the third group with funded updates. For all groups, no additional blood samples will be drawn for research purposes; only routinely obtained clinical data will be used. The primary outcome in all groups will be the percentage of participants with appropriate vancomycin concentrations. Secondary outcomes in those who receive vancomycin for at least 72 hours will include effectiveness, toxicity rates, and costs of therapy. Participation in the study will cease at the time of hospital discharge or 72 hours after termination of vancomycin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized infants, children, adolescents, and adults who require, but have not started vancomycin therapy for infections with suspected or proven beta-lactam resistant gram-positive bacteria will eligible for enrollment.
2. Participants will of any age.
3. Participant/parent/legal guardian (as applicable) must be able and willing to provide signed informed consent.

Exclusion Criteria:

1. Prior receipt of vancomycin for the same clinical event (e.g. the same fever of unknown origin in a neutropenic patient defined as <24 hours of no fever)
2. Known colonization or infection with a vancomycin resistant organism (MIC > 2 mg/L)
3. Known hypersensitivity or intolerance to vancomycin
4. Patients on any form of dialysis
5. Not expected to survive >72 hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized infants, children, adolescents, and adults who require, but have not started vancomycin therapy for infections with suspected or proven beta-lactam resistant gram-positive bacteria will eligible for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-04 (Actual)

PRIMARY OUTCOMES:
Time to therapeutic vancomycin blood concentration | Within first week of dosing

SECONDARY OUTCOMES:
Number of blood samples sent for vancomycin concentration measurement | Duration of therapy, an average of 10 days in the hospital
Incidence of nephrotoxicity | Duration of therapy, an average of 10 days in the hospital
  Defined as >0.5 mg/dL or >50% rise from baseline serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Michael Neely, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Los Angeles County - University of Southern California Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual data requests will be evaluated on a case-by-case basis.

REFERENCES:
- [Derived] Neely MN, Kato L, Youn G, Kraler L, Bayard D, van Guilder M, Schumitzky A, Yamada W, Jones B, Minejima E. Prospective Trial on the Use of Trough Concentration versus Area under the Curve To Determine Therapeutic Vancomycin Dosing. Antimicrob Agents Chemother. 2018 Jan 25;62(2):e02042-17. doi: 10.1128/AAC.02042-17. Print 2018 Feb. PMID 29203493